CLINICAL TRIAL: NCT05680558
Title: THERAKOS® CELLEX Photopheresis System as an Interventional Therapy for the Treatment of Early Stage CTCL (Mycosis Fungoides), an Open-label, Single-arm, Multi-center, Phase II Study
Brief Title: Photopheresis in Early-stage Mycosis Fungoides
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Mallinckrodt, Inc. (Unknown)
Responsible Party: Principal Investigator, Larisa Geskin, MD, Director, Cutaneous Oncology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS9960
Record Dates: First submitted 2022-11-12; First posted 2023-01-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cutaneous T Cell Lymphoma; Mycosis Fungoides
Keywords: photopheresis
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- UVA Sterile Solution in conjunction with the THERAKOS® CELLEX Photopheresis System (Experimental): TREATMENT with THERAKOS® CELLEX Photopheresis System on two consecutive days every 2 weeks for the first 3 months; then once per month for following 9 months.
  Interventions: Drug: UVADEX® (methoxsalen) Sterile Solution in conjunction with the THERAKOS® CELLEX Photopheresis; Device: THERAKOS® CELLEX photopheresis system

INTERVENTIONS:
Drug: UVADEX® (methoxsalen) Sterile Solution in conjunction with the THERAKOS® CELLEX Photopheresis — Extracorporeal Photopheresis (ECP)
  Other Names: UVADEX® with THERAKOS® CELLEX Photopheresis
Device: THERAKOS® CELLEX photopheresis system — THERAKOS® CELLEX is an FDA-approved extra-corporeal photopheresis system

SUMMARY:
The purpose of this study is to determine whether photopheresis therapy can be used to improve the clinical course of early stage cutaneous T-cell lymphoma (CTCL). Currently, photopheresis is performed as a palliative treatment for late stage CTCL. However, recent studies have demonstrated that patients with early stage CTCL may have markers in their blood which were previously observed primarily in late stage disease, such as clonal T cell populations. Considering these findings, the study aims to investigate whether photopheresis therapy may be used earlier in the disease course to produce a clinical response.

DETAILED DESCRIPTION:
The THERAKOS® CELLEX Photopheresis System is currently FDA approved and indicated for the palliative treatment of the skin manifestations of cutaneous T-cell lymphoma (CTCL) in patients not responsive to other forms of treatment. The original studies in CTCL were performed in patients having extensive patch/plaque or erythrodermic stage disease. Therefore, photopheresis is used primarily to treat stage III or IV CTCL. However, studies have shown that 50% of patients with early disease may have clonal T-cells in their peripheral blood if polymerase chain reaction is used to amplify the T-cell receptor gamma gene fragments. Thus, patients who are staged as T1 or T2 who also have slight abnormalities in blood involvement, such as atypical cells seen on blood smear or abnormal flow cytometry may benefit from photopheresis therapy. This study aims to investigate the efficacy of photopheresis therapy in patients with Stage !A, 1B, or IIA CTCL.

ELIGIBILITY:
Inclusion Criteria:

1. Who are male or female, over the age of 18 and <40 kg body weight with adequate veins to provide intravenous access.
2. Who are willing to adhere to the protocol and sign an Informed Patient Consent Document
3. Must not be on any other investigational device/drug treatment.
4. Who have the diagnosis of Mycosis Fungoides (MF) including a skin biopsy consistent with MF (atypical epidermotropic or folliculocentric T-cells) with appropriate staging as IA, IB or IIA: T1 or T2 (patches or plaques) with measurable lesions.
5. With IA stage must demonstrate a minor blood abnormality by morphology/laboratory assessment.
6. With IIA stage - clinically significant nodes (1.5 cm) must have lymph node biopsy showing dermatopathic nodes or no involvement.
7. Must be willing and able to discontinue concomitant medications for MF. Subjects currently taking the following drugs must discontinue medication with the following wash out periods prior to enrollment in the trial: PUVA or UVB Therapy - 4 weeks, topical nitrogen mustard or other topical chemotherapy - 4 weeks, bexarotene capsules or other systemic biologic agent - 3 weeks washout, high dose topical steroids, topical retinoids or immunotherapy - 2 week washout with 1% topical hydrocortisone , oral steroids above 10 mg - 30 day washout, unless subject has Addison's Disease or adrenal insufficiency
8. Who are refractory to at least one of the standard therapies used to treat Stage IA, IB or IIA CTCL such as oral steroids, high-dose topical steroids, topical nitrogen mustard, Bexarotene, PUVA therapy, electron beam radiation, biological response modifiers or oral methotrexate.
9. Must be willing to abstain from therapeutic sunbathing, phototherapy, tanning beds, etc. for the duration of the study.

Exclusion Criteria:

1. Who have MF (T3 cutaneous tumors or T4 exfoliative erythroderma) Stage IIB - IVB
2. Who are unable to tolerate extracorporeal volume loss i.e., severe cardiac disease/anemia
3. With deterioration of renal function who have a serum creatinine level greater than 3.0 mg/dL.
4. With lipemic plasma >500 ng/dL, uncontrolled diabetes, history of liver damage (2.5 x normal alanine transaminase (ALT), aspartate aminotransferase (AST), porphyria, lupus, positive tests for human immunodeficiency virus (HIV) antibody, hepatitis C virus (HCV) antibody or Hepatitis B Surface Antigen, severe emotional, behavioral or psychiatric problems that, in the opinion of the investigator, would result in poor compliance with the treatment regimen, and idiosyncratic or hypersensitivity reactions to 8-methoxypsoralen compounds, heparin, or citrate.
5. On oral prednisone therapy or high potency topical steroids.
6. Who are pregnant or nursing a child.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-05-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 1 Year
  Overall response rate at 1 year measured by the modified skin-weighted assessment tool (mSWAT) in accordance with Olsen et al criteria for response in clinical trial. Measurable lesions are defined as those that can be accurately measured in at least one dimension.

SECONDARY OUTCOMES:
Time to Response of Photopheresis Therapy | 1 Year
  The time to response calculated from time of photopheresis treatment initiation to the first objective response (clearance of skin disease from baseline ≥50%) observed for participants who achieved a complete response (CR) (clearing of all disease manifestations confirmed by biopsy) or partial response (PR) (partial response defined as > 50% improvement in the extent of skin involvement).
Duration of Response | 1 Year
  Duration of response (DOR) will be calculated from time of response to documentation of progression or death.
Change in Functional Assessment of Cancer Therapy - General (FACT-G) Score | Baseline and 1 Year
  The FACT-G is a 27-item questionnaire designed to measure four health related quality of life in cancer patients. Scores range from 0-108 with a higher score indicating better quality of life.
Change in Skindex-29 Score | Baseline and 1 Year
  The Skindex-29 is a questionnaire with 29 questions that assess the health-related quality of life of patients with skin diseases. Scores range from 0-100 with a higher scoring indicating a worse health status.
Change in Short Form Survey (SF-36v2) Score | Baseline and 1 Year
  The SF-36v2 is a health survey measuring quality of life. Scores range from 0-100 with a higher scoring indicating a better quality of life.
Change in Size of Lymph Nodes | Baseline and 1 Year
  The change in size (single maximum dimension in centimeters) of lymph nodes will be noted as applicable. By definition, the patients should not have pathologically involved lymph nodes.
Change in Sézary Cell Counts at 6 and at 12 months | Baseline, 6 months and 12 months
  Change in Sézary cell counts (malignant cells) in blood samples as assessed by flow cytometry. By definition, the enrolled patients will have only minor blood involvement and not leukemia.

CONTACTS AND LOCATIONS:
Overall Officials: Larisa Geskin, MD, Principal Investigator — Columbia University
Locations (1):
- Herbert Irving Pavilion, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No